CLINICAL TRIAL: NCT02245698
Title: Autologous Bone Marrow Mononuclear Cells Intrathecal Transplantation in Stroke
Brief Title: Autologous Stem Cell Therapy in Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-11
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: Chronic Stroke; Subacute stroke; Autologous Bone Marrow Mononuclear Cell therapy; Stem cell
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): Bone marrow mononuclear cells
  Interventions: Biological: Stem cell

INTERVENTIONS:
Biological: Stem cell — Intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to study the safety and effect of stem cell therapy on the functional recovery in patients with sub acute/chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age18 years-80 years
* diagnosed as stroke by clinical and MRI findings

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/ Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever
* hemoglobin less than 8
* bleeding tendency
* bone marrow disorder
* left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure | 1 year
  Functional Independence Measure scale assesses the patients ability to carry out activities of daily living. At the follow up of 1 year, every patient in this study will be reevaluated on this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided